CLINICAL TRIAL: NCT00694434
Title: Graduated Embryo Score (GES) Int he Fresh Cycle Predicts Outcome From Frozen Embryo Transfer
Brief Title: Graduated Embryo Score (GES) in the Fresh Cycle Predicts Outcome From Frozen Embryo Transfer
Acronym: GES/FET
Status: Completed | Type: Observational
Sponsor: Sher Institute for Reproductive Medicine, Las Vegas (Other)
Responsible Party: Jeffrey Fisch, M.D., Sher Institute
Other Study IDs: 1-Fisch
Record Dates: First submitted 2008-06-06; First posted 2008-06-10 (Estimated); Last update posted 2008-06-10 (Estimated); Status verified 2008-06

CONDITIONS: Infertility
Keywords: Cryopreservation; Frozen embryo transfer; Graduated Embryo Score
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients with 2 or more frozen blastocyst that scored GES 70 or better in the fresh cycle.
- 2: Patients with 2 or more frozen blastocysts scoring GES <70 in the fresh cycle.

SUMMARY:
Evaluation of embryo quality in the fresh cycle as a predictor of outcome from frozen embryo transfer.

DETAILED DESCRIPTION:
Outcomes from frozen embryo transfer reviewed based on the quality of the embryos in the ftresh cycle as assessed by the Graduatede embryo score.

ELIGIBILITY:
Inclusion Criteria:

* 2 frozen blastocysts

Ages: 21 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All IVF patients at our center between 2002 and 2007 with at least 2 frozen blastocysts undergoing frozen embryo transfer.
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2002-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
On-going gestation (beyond 8 wks) | Fetal heart activity at 8 weeks of gestation

SECONDARY OUTCOMES:
Implantation rate (gestational sacs/ embryos transferred) | 8 weeks of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey D Fisch, M.D., Principal Investigator — Sher Institute
Locations (1):
- Sher Institute for Reproductive Medicine, Las Vegas, Nevada, United States